CLINICAL TRIAL: NCT03155360
Title: Association Between Infant Colics and Parental Migraine ? Non Interventional Study in the Pediatric Emergency Unit of Nancy (France) University Hospital
Brief Title: Infants Colics : Towards a Migrainous Origin ?
Acronym: COLIGRAINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00185-48
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Colic, Infantile; Migraine; Migraine Equivalents
Keywords: Colics; infant colics; Migraine equivalent; Migraine; Episodic symptoms associated to migraine; Colic
MeSH Terms: conditions — Colic; Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infant with colics: Infants with colics according to Wessel definition :
  * Recurrent episodes of irritability, fussing or crying from birth to 4 months of age
  * Episodes last for 3 hours per day ; on 3 days per week ; for 3 weeks
  * Episodes can not be attributed to another disorder
  Interventions: Other: Non interventional study
- Infant without colics
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Non interventional study

SUMMARY:
According to recent studies, we want to find evidences that infant colics could be a episodic symptom associated to migraine as cyclic vomiting syndrome or abdominal migraine are. The main purpose is to compare the presence of colics in infants between 60 days and 180 days of life and the presence of migraine in their parents to determine if colicky children's parents are more migrainous than other parents.

DETAILED DESCRIPTION:
Recent studies shows that :

* Infants with colics have more probability to become migrainous when they will grow up
* Migrainous children have more colic history in their past
* Migrainous parents have more babies with colics than non-migrainous parents

According to these studies, we want to find othen evidences that infant colics could be a migraine equivalent as cyclic vomiting syndrome or abdominal migraine are. Recently, the international classification of headache disease IIIbeta added in its appendix colics in the episodic symptoms associated to migraine

The main purpose of our study in the pediatric emergency unit of Nancy is to compare the presence of colics in infants and the presence of migraine in their parents to determine if colicky children's parents are more migrainous than other parents. The data collection will be made thanks to a survey which will be completed by the parents.

ELIGIBILITY:
Inclusion Criteria:

* All infants between 60 days and 180 days of life who comes to the Nancy University Hospital pediatric emergency unit

Exclusion Criteria:

* Language barrier of parents

Ages: 60 Days to 180 Days | Sex: All
Age Groups: Child
Study Population: All infants between 60 days and 180 days of life who comes to the Nancy University Hospital pediatric emergency unit
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of real colics according to Wessel definition | At the inclusion
Proportion of migrainous parents | At the inclusion
  Proportion of migrainous parents in each group

SECONDARY OUTCOMES:
Proportion of Infant colics according the feeling parents | At the inclusion
Proportion of maternal migraine | At the inclusion
Proportion of partenal migraine | At the inclusion
Age of begining of colics | At the inclusion
  average and median age
Age of ending of colics | At the inclusion
  average and median age
Proportion of real colics according to Wessel definition in the subgroup of parents who report that their child has colic | at the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Dr BORSA-DORION Anne, Nancy, France

IPD SHARING:
Plan to Share IPD: No